CLINICAL TRIAL: NCT03196869
Title: Phase II Clinical Randomized Study of the Effect of Chronomodulated Chemotherapy Followed by Concurrent IMRT Chemo-radiotherapy on the Dendritic Cells Subsets and Immunity in the Treatment of Advanced Nasopharyngeal Cancer
Brief Title: the Study of Effect of Chronomodulated Chemotherapy on the Dendritic Cells Subsets in the Treatment of Advanced Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201708112121
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: NPC peripheral blood dendritic cell chronic-chemotherap
MeSH Terms: interventions — Control Groups; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chrono-chemotherapy group (Experimental): Induction chrono-chemotherapy followed by cisplatin chrono-chemotherapy concurrent combined with intensity-modulated radiation therapy;Delivery time is different from the control group
  Interventions: Device: Chrono-chemotherapy; Drug: induction Chrono-chemotherapy; Drug: cisplatin chrono-chemotherapy; Radiation: intensity-modulated radiation therapy
- Routine intravenous drip (Other): control group:Induction routine-chemotherapy followed by cisplatin routine-chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Device: Routine intravenous drip; Drug: induction Routine-chemotherapy; Drug: cisplatin routine-chemotherapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Device: Chrono-chemotherapy — Chrono-chemotherapy+concurrent radiochemotherapy
  Other Names: Experimental group
  Arms: Chrono-chemotherapy group
Device: Routine intravenous drip — Routine intravenous drip-chemotherap
  Other Names: control group
  Arms: Routine intravenous drip
Drug: induction Chrono-chemotherapy — Experimental group:docetaxel,cisplatin,5-FU
  Other Names: chronological dosage
  Arms: Chrono-chemotherapy group
Drug: induction Routine-chemotherapy — control group:docetaxel,cisplatin,5-FU
  Other Names: Conventional drug delivery
  Arms: Routine intravenous drip
Drug: cisplatin chrono-chemotherapy — Experimental group: cisplatin chrono-chemotherapy
  Other Names: cisplatin Conventional drug delivery
  Arms: Chrono-chemotherapy group
Drug: cisplatin routine-chemotherapy — control group:cisplatin routine-chemotherapy
  Other Names: cisplatin Conventional drug delivery
  Arms: Routine intravenous drip
Radiation: intensity-modulated radiation therapy — control group is similar to Experimental group

SUMMARY:
This study is to observe and compare the effect of docetaxel plus lobaplatin induction chemotherapy combined with lopoplatin chemoradiotherapy and TPF induction chemotherapy combined with cisplatin chemoradiotherapy on dendritic cells subsets in the treatment of locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
TPF program is currently the local advanced head and neck squamous cell carcinoma commonly used inducing chemotherapy, cisplatin is the preferred drug for the same period chemotherapy.Dendritic cells (DC) play an essential role in the induction and regulation of immune responses.The effect of radiation and chemotherapy is closely related to the patients' immune function.In this study, Phase II clinical trials were performed. Patients with locally advanced head and neck squamous cell carcinoma were randomly divided into experimental group and control group. The trial group was treated with docetaxel + lorosine-induced chemotherapy combined with lorplatin concurrent radiotherapy and chemotherapy. The control group was treated with TPF Cisplatin concurrent chemotherapy, observed the relationship between dendritic cells subsets and clinical prognosis of patients, to provide a new method for the treatment of locally advanced nasopharyngeal carcinoma and technical support

ELIGIBILITY:
Inclusion Criteria:

1. initial treatment of advanced nasopharyngeal carcinoma Ⅲ-Ⅳ patients with pathologically confirmed (according to 2010 UICC staging, T3-4, N0-3), without evidence of distant metastasis (M0). Have measurable tumor lesions.
2. KPS≥70 points.
3. the age of 18-70 years old, male or female.
4. no major organ dysfunction; normal bone marrow function (WBC ≥4.0 × 109 / L, platelets ≥100 × 109 / L, hemoglobin ≥90g / L), normal liver function (total bilirubin, alanine aminotransferase, aspartate aminotransferase ≤1.5 times the upper limit of normal), normal renal function (creatinine ≤ 1.5 times upper limit of normal).
5. understand this study and signed informed consent

Exclusion Criteria:

1. Three months in the use of Chinese herbal medicine or immune modulators
2. distant metastasis.
3. who had received prior chemotherapy.
4. patients have physical or mental illness, and by researchers believe that patients can not be completely or fully understood in this study possible complications.
5. pregnancy (via the urine or serum β-HCG test confirmed) or during lactation. serious complications, such as uncontrolled hypertension, heart failure, diabetes and so on.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-04-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Dendritic cell subgroup changes of Participants | termination of treatment, 3 months after treatment
  By flow cytometry detection of two groups of peripheral blood dendritic cells subsets and lymphocyte subpopulation changes before and after the radiation and chemotherapy

SECONDARY OUTCOMES:
Number of Participants with curative effect | 1 year
  Evaluate the immediate effect at 1year after Concurrent chemo-radiotherapy by RECIST
Number of Participants with Adverse Events as a Measure of Safety | 5 year
  To assess and record nausea, vomiting, oral mucositis, diarrhea and other adverse drug reactions by CTC 4.0

OTHER OUTCOMES:
Progression-free survival | 5 years
  Evaluate the Progression-free survival at five years after Concurrent chemo-radiotherapy by RECIST.
Overall survival | 5 years
  Evaluate the Overall survival at five years after Concurrent chemo-radiotherapy by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jin, Bachelor, Study Chair — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No